CLINICAL TRIAL: NCT05482698
Title: A Parallel-group (2-Arm), Randomized, Double-blind, 12-week Trial to Evaluate the Efficacy and Safety of MC2-25 Cream and MC2-25 Vehicle in Subjects With Chronic Kidney Disease-associated Pruritus (CKD-aP)
Brief Title: The MC2-25 Cream in Subjects wITh CHronic KIdNEy Disease-aSsociated prurituS (ITCHINESS) Trial
Acronym: ITCHINESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MC2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MC2-25-C1
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Results first posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Chronic Kidney Disease-associated Pruritus

STUDY DESIGN:
Intervention Model Description: Parallel-group, Randomized, Double-blind
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MC2-25 cream (Experimental): MC2-25 cream Twice daily applications for 12 weeks
  Interventions: Drug: MC2-25 cream
- MC2-25 vehicle (Placebo Comparator): MC2-25 vehicle Twice daily applications for 12 weeks
  Interventions: Drug: MC2-25 vehicle

INTERVENTIONS:
Drug: MC2-25 cream — Topical application
  Arms: MC2-25 cream
Drug: MC2-25 vehicle — Topical application
  Arms: MC2-25 vehicle

SUMMARY:
The purpose of this study is to access the efficacy and safety of MC2-25 cream and MC2-25 vehicle for treatment of chronic kidney disease associated pruritus (CKD)-aP).

DETAILED DESCRIPTION:
In this trial, subjects who fulfil all inclusion and exclusion criteria are enrolled.

Eligible subjects will be randomised in a 2:1 ratio to MC2-25 cream or MC2-25 vehicle, respectively.

The subjects will apply the assigned investigational medicinal product (IMP) twice daily for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or non-pregnant females of any race or ethnicity who are ≥ 18 years of age at the time of screening
* Has provided written informed consent
* Chronic (>3 months) kidney disease (CKD) stages G3-G5 (i.e., estimated glomerular filtration rate [eGFR] by CKD-EPI creatinine 2021 equation <60 mL/min/1.73 m2)
* Specifically for CKD subjects on haemodialysis (HD) or haemodiafiltration (HDF):

  1. Subjects must be established on HD or HDF 3 times per week continuously for at least 3 months prior to the start of screening and must not have plans to change from HD to HDF or vice versa during the trial
  2. Subjects who require an occasional additional HD or HDF treatment to manage fluid overload may be enrolled as long as it is anticipated that no more than 4 such treatments will be required in any given month
* At least moderate CKD-aP defined as WI-NRS ≥4
* Female subjects must be of either: a. Non-childbearing potential or b. Childbearing potential

Exclusion Criteria:

* Has a functioning kidney transplant or is scheduled to receive a kidney transplant during the trial (Note: subject can be on waiting list for kidney transplant)
* Subjects who receive peritoneal dialysis
* In the opinion of the investigator has pruritus attributed to a cause other than CKD or its complications
* Has localized itch restricted to the palms of the hands
* Has concurrent skin conditions (including but not limited to pruritic dermatoses, active skin infections, ulcerations) that may limit or prevent application of MC2-25 cream or MC2-25 vehicle or that may interfere with evaluation of the effects of MC2-25 cream or MC2-25 vehicle on the skin at the Screening or Baseline visits
* Subjects who will have skin biopsies performed must not have any known hypersensitivity to the local anaesthetic or diagnosed bleeding disorders
* Has a concurrent or recent (within 12 months prior to screening) medical condition that, in the opinion of the investigator, could pose undue risk to the subject, impede completion of the trial procedures, or would compromise the validity of the trial measurements
* Has a known current generalized infection (bacterial, viral, or fungal)
* Start of a new or change to existing systemic treatment for CKD-aP
* Use of emollients on CKD-aP areas within 10 days prior to the Baseline visit
* Use of any topical treatment on CKD-aP areas
* Use of any light therapy for CKD-aP
* Use of non-biologic systemic immunosuppressive treatment
* Use of biologic systemic treatment
* Subjects not currently on dialysis but who are likely to initiate routine dialysis during participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MC2-25 Cream | MC2-25 Vehicle
Started | 73 | 38
Completed | 65 | 33
Not Completed | 8 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MC2-25 Cream | MC2-25 Vehicle | Total
Number analyzed (Participants) | 73 | 38 | 111
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.0 (15.13) | 66.9 (13.78) | 63.7 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 16 | 53
  Male | 36 | 22 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 73 | 38 | 111
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 5 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 1 | 7
  White | 55 | 31 | 86
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 41 | 22 | 63
  Germany | 10 | 6 | 16
  Hungary | 22 | 9 | 31
  Poland | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Weekly Mean Worst Itch Numeric Rating Score (WI-NRS)
Description: Mean change in WI-NRS score, calculated as the average of weekly means WI-NRS values from Baseline to Week 12 for MC2-25 cream compared to MC2-25 vehicle. Weekly mean WI-NRS is calculated as the average of all and at least 4 non-missing WI-NRS values recorded in the subjects' diaries for the 7 days prior to and including the scheduled in clinic visits (8 days in total expected). The WI-NRS was scored on a 11-point numeric rating scale ranging from 0 to 10, where 0=no itch and 10=worst imaginable itch.
Time Frame: 12 weeks
Population: The number (59/34) of participants in the full analysis set is the number of subjects with at least a baseline weekly mean WI-NRS score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MC2-25 Cream | MC2-25 Vehicle
Number analyzed (Participants) | 59 | 34
score on a scale | -3.70 (2.961) | -3.87 (2.203)

ADVERSE EVENTS:
Time Frame: Adverse event information was collected from individual trial subjects from signature of the informed consent form and through study completion, i.e. for a maximum of 18 weeks.
Arm/Group | MC2-25 Cream | MC2-25 Vehicle
All-Cause Mortality (participants affected / at risk) | 1/73 | 1/37
Serious Adverse Events (participants affected / at risk) | 11/73 | 6/37
Other Adverse Events (participants affected / at risk) | 4/73 | 2/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC2-25 Cream (N=73) | MC2-25 Vehicle (N=37)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Hematomas in the area of the left elbow joint and the laft knee joint (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC2-25 Cream (N=73) | MC2-25 Vehicle (N=37)
Application site pain (General disorders) | 4 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT05482698/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT05482698/SAP_001.pdf